CLINICAL TRIAL: NCT04216862
Title: Effect of Strengthening and Stretching Exercise of Deep Neck Muscles Group to Improve Forward Head Posture and Rounded Shoulders in Normal Healthy Adults
Brief Title: Strengthening and Stretching Exercise to Improve Forward Head Posture and Rounded Shoulders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Tehmina Irfan
Record Dates: First submitted 2019-12-23; First posted 2020-01-03 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Forward Head Posture
Keywords: Forward Head; Rounded Shoulder; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening exercise treatment (Experimental): This exercise targets the deep flexor muscles of the upper cervical region the longus capitis and longus colli muscles.
  Interventions: Other: Exercise
- Stretching exercise treatment (Active Comparator): The subject's forearm is stabilized by a vertical plane before the trunk is rotated in the opposite direction. Therefore the arm on the involved side is externally rotated and abducted to 90.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Different type of exercises for treatment of Forward Head Posture

SUMMARY:
Forward head posture (FHP) and Rounded shoulders (RS) are defined as protrusion of the head and shoulders in the sagittal plane. Forward head posture is defined as the anterior positioning of the cervical spine. Rounded shoulders also called protracted shoulder (PS) is a protrusion of the acromion of the shoulder joint relative to the centerline of gravity of the body, causing stooped posture along with elevation, protraction, and downward rotation of the scapula, and an increased angle between the lower neck bone and upper spine. Many Physical therapy treatment options are available to correct forward head posture and rounded shoulders which focused to correct the muscle imbalance and restore the normal posture of Cervical spine and shoulder. The objective of this study is to compare the outcomes of Strengthening exercise with the outcomes of stretching exercise on the targeted muscle group to correct forward head posture and rounded shoulders. The study will determine effective management plan for correction of forward head posture and rounded shoulders. It will be Experimental Randomized Controlled Trial. 26 Patients will be included through consecutive sampling, with 13 patients in each of 2 groups. Subjects will be equally distributed to two groups with use of dice roll method of randomization. From the two groups, one receiving strengthening exercise treatment and other receiving stretching exercise treatment. Statistical Package for Social Sciences (SPSS) V 25.will be used for Data analysis. Results will be extracted. Conclusion will be made after comparing the pre and post treatment results of both treatment approaches.

DETAILED DESCRIPTION:
Forward head posture and Rounded Shoulder are related to muscle imbalance, which disturbs length tension relationship of muscles. Weak and lengthened muscles in Forward head posture and rounded shoulders are deep neck flexors which include longus capitis and longus coli and weak scapular stabilizers and retractors which include Rhomboids and middle, lower trapezius, Teres Minor and Infraspinatus. The overactive and shortened muscles participating in Forward head posture and Rounded shoulders are Deep upper cervical extensors which include longissimus capitis, Splenius Capitis, Cervical Multifidus, Upper Trapezius and Shoulder protractors and elevators which include Pectoralis minor, Pectoralis major and Levator Scapula. Previous researches suggests that weakened postural muscles should be strengthened and shortened muscles should be lengthened in order to improve postural alignment and alleviate Forward head posture and restoring the normal muscle balance between opposing muscle groups (agonists and antagonists). The majority of treatments have focused on the deep neck flexors, as they play a major role in stabilizing the alignment of the cervical spine. Exercise improved the forward head and Rounded Shoulder significantly.

The selection of 50º as a reference angle for forward head posture was guided by previous studies, with the latter reporting 55.02 ± 2.86 as a normal range. As is well known, subjects with forward head posture have a significantly smaller cervical angle when compared with normal subjects. In the present study, the investigators considered 52º as the reference angle based on a previous study which evaluated 310 participants in a standing position and reported 2.6º±15.3 as a normal range, and Brink et al, who evaluated 15 to 17 year-olds and reported a mean shoulder angle value of 51.35º ± 17.2º, and based on the premise that subjects with protracted shoulder have a significantly smaller shoulder angle when compared with normal subjects. Individual will be considered to have rounded shoulder if the angle will be less than 52º.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals having Craniovertebral Angle (CVA) less than 50 degree
2. Individuals having Shoulder Angle (SA) less than 52 degree.
3. Those who had not under any regular exercise for last 6 months
4. Those who use a smart phone or computer for at least 4 hours or more per day on average.

Exclusion Criteria:

1. Individuals will be excluded if they had visual deficits, diagnosed balance disorders, musculoskeletal pathologies (e.g. history of shoulder surgery, cervical or thoracic fracture, Osteosarcoma, Myeloma), non-ambulatory, displayed functional or structural scoliosis, or had excessive thoracic kyphosis.
2. Individuals having symptoms of Vertebral Artery Insufficiency.
3. Individuals not willing to participate or to follow up treatment plan.

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Craniovertebral angle | 3 Months
  The angle between the line from the external auditory meatus to the seventh cervical vertebra and a horizontal line at the level of the seventh cervical vertebra using photogrammetry
Scapular Index | 3 Months
  Its the ratio of the length of the scapula to its breadth multiplied by 100 and will be measured using Posture Assessment Software

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynch SS, Thigpen CA, Mihalik JP, Prentice WE, Padua D. The effects of an exercise intervention on forward head and rounded shoulder postures in elite swimmers. Br J Sports Med. 2010 Apr;44(5):376-81. doi: 10.1136/bjsm.2009.066837. PMID 20371564
- [Background] Lee MH, Park SJ, Kim JS. Effects of neck exercise on high-school students' neck-shoulder posture. J Phys Ther Sci. 2013 May;25(5):571-4. doi: 10.1589/jpts.25.571. Epub 2013 Jun 29. PMID 24259804
- [Background] Lee DY, Nam CW, Sung YB, Kim K, Lee HY. Changes in rounded shoulder posture and forward head posture according to exercise methods. J Phys Ther Sci. 2017 Oct;29(10):1824-1827. doi: 10.1589/jpts.29.1824. Epub 2017 Oct 21. PMID 29184298
- [Background] Diab AA, Moustafa IM. The efficacy of forward head correction on nerve root function and pain in cervical spondylotic radiculopathy: a randomized trial. Clin Rehabil. 2012 Apr;26(4):351-61. doi: 10.1177/0269215511419536. Epub 2011 Sep 21. PMID 21937526
- [Background] Falla D, Jull G, O'Leary S, Dall'Alba P. Further evaluation of an EMG technique for assessment of the deep cervical flexor muscles. J Electromyogr Kinesiol. 2006 Dec;16(6):621-8. doi: 10.1016/j.jelekin.2005.10.003. Epub 2005 Dec 15. PMID 16359872